CLINICAL TRIAL: NCT01834599
Title: Could the Cerebral Oximetry (NIRS) be a Good Technology to Measure Placental Oxygenation in Pregnant Woman?
Brief Title: Could the Cerebral Oximetry be a Good Technology to Measure Placental Oxygenation?
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Christian Loubert, Christian Loubert, MD, FRCPC, Maisonneuve-Rosemont Hospital
Other Study IDs: LoubertHMR2013/04
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Placental Oxygenation
Keywords: placental oxygenation; obstetric anesthesia; NIRS; cerebral oximetry; cerebral oximeter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- anterior placenta: Cerebral oximetry device used to obtain:
  Saturation value of the placenta probe with no oxygen, saturation value of the placenta probe with oxygen, saturation value of the myometrium probe with no oxygen saturation value of the myometrium probe with oxygen saturation value of the forearm probe with no oxygen, saturation value of the forearm probe with oxygen saturation value of the leg probe with no oxygen saturation value of the leg probe with oxygen Timing between the contractions measure by cardiotocography
  Interventions: Device: cerebral oximetry

INTERVENTIONS:
Device: cerebral oximetry — tissue saturation measurement in pregnant women
  Other Names: NIRS; INVOS

SUMMARY:
To assess the potential of the cerebral oximeter to measure placental oxygenation

DETAILED DESCRIPTION:
There is general agreement among experts to recommend the use of phenylephrine as first line therapy for the treatment of arterial hypotension induced by spinal anaesthesia during caesarean delivery. In some studies, there are trends toward a lower PaO2 values in the umbilical cord venous blood when the mother receive this vasopressor. These findings may be a result of the vasoconstrictor effect of phenylephrine on utero-placental vessels, and a subsequent increased oxygen extraction by the fetus. The possibility to extract more oxygen would provide a certain "safety margin" in the event of compromised utero-placental blood flow during normal pregnancy. However, this "safety margin" should not be taken for granted in cases where signs of fetal distress are present, and this situation might influence the choice of vasopressors.

It is well establish on a physiological basis that during labour, utero-placental blood flow is lower during the contractions. This lower blood flow could result in a lower saturation value measured by the cerebral oximeter.

Twenty patients in labour will be included in this study. Patients will be recruited in obstetric clinic during pregnancy. Based on the second trimester ultrasound, patients with anterior placenta will be included.

During labour, once a functional epidural is in place, an Invos oximeter will be install. Two sensors will be applied on the abdomen (one above the placenta and the other above the myometrium at a place without placenta). Two sensors will also be applied on the extremities (forearm and leg).Saturation values and timing of the contractions will be recorded for sixty minutes. Half of the recording will be done with an oxygen mask. Vitals signs will also be registered every five minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant woman (ASA I or II)
* Term gestation ( > 37 weeks)
* Normal pregnancy
* vaginal delivery
* obstetrical epidural in place
* anterior placenta

Exclusion Criteria:

* patient refusal
* Any contraindication to neuraxial anesthesia
* cesarean section
* multiple gestation
* placentation abnormalities
* anormal placental perfusion
* Placental Abruption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: healthy pregnant woman at term gestation in labour
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference between Δp and Δm | 60 minutes
  Δp = Difference between the mean value area under the curve for the placenta and arm = (Ap- Af) Δm= Difference between the mean value area under the curve for the myometrium and arm = (Am- Af)

SECONDARY OUTCOMES:
Difference of the area under the curve of saturation with and without oxygen | 60 minutes
  Ap with Oxygen - Ap without oxygen; Am with oxygen - Am without oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Christian Loubert, MD, FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada